CLINICAL TRIAL: NCT01415973
Title: Nutrient Synergy in Beef and Stimulation of Protein Synthesis in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UAMS IRB #132559
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: beef; protein; synergy; intact beef constituents; protein constituent; Nutrient Synergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 ounces of cooked, 85% lean ground beef (Experimental): Subjects would consume 3 ounces of cooked, 85% lean ground beef at one setting on one day.
  Interventions: Dietary Supplement: 3 ounces of cooked, 85% lean ground beef
- 20 grams of Beef protein isolate (Experimental): Subjects would consume 20 grams of beef protein isolate dissolved into 200mL water at one setting on one day.
  Interventions: Dietary Supplement: 20 grams beef protein isolate

INTERVENTIONS:
Dietary Supplement: 3 ounces of cooked, 85% lean ground beef — Consumed once per subject.
  Arms: 3 ounces of cooked, 85% lean ground beef
Dietary Supplement: 20 grams beef protein isolate — Subjects would drink 200 ml water mixed with 20 grams of beef protein isolate one time.
  Arms: 20 grams of Beef protein isolate

SUMMARY:
This study will compare the effects of cooked, ground beef to those of beef protein isolate on blood and muscle proteins.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Primary: To compare the effects of consumption of a 3-ounce serving of beef to that of a 20g serving of BPI on skeletal muscle synthetic and breakdown rate in healthy elderly subjects.

Secondary: To investigate the effect the study products on plasma levels of amino acids, insulin, and glucose in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female.
* Age 60 years or older.

Exclusion Criteria:

* Any (history of) gastrointestinal disease that interferes with GI function
* Diagnosed and active treatment of Diabetes Mellitus type I or II
* History of congestive heart failure
* Recent (6 months) hospitalization for heart disease treatment or management (e.g. PTCA, stent, surgery)
* Myocardial infarction in the past year
* Infection or fever in the 7 days prior to enrollment
* Current use of corticosteroids, growth hormone, or testosterone
* Adherence to a weight loss diet
* Use of protein-containing or amino acid-containing nutritional supplements within one week of enrollment
* Current alcohol (>7 ETOH per week) or drug abuse
* Platelet count (PLT) < 100,000
* History of hypo- or hyper-coagulation disorders including use of a coumadin derivative
* Currently taking anti-thrombotics and cannot stop for 7 days (i.e. medical indication)
* Allergy to local anesthetic
* Blood hemoglobin < 9.0 g/dL
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
skeletal muscle synthetic and breakdown rate | day one
  Using stable isotope infusion/ingestion methodology, we will measure plasma and skeletal muscle metabolic rate. Our primary end points will be muscle protein fractional synthesis rate (FSR) and whole body protein turnover rate.

SECONDARY OUTCOMES:
concentrations of plasma amino acids, insulin and glucose | day one
  Secondary endpoints are concentrations of plasma amino acids, insulin and glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Wolfe, PhD, Principal Investigator — UAMS
Locations (1):
- UAMS Center on Aging, Little Rock, Arkansas, United States